CLINICAL TRIAL: NCT00581841
Title: Repeatability of X-Ray, MRI, and Gait Analysis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Kenton R. Kaufman, PhD, PE, Mayo Clinic
Other Study IDs: R01 AR48768 - substudy; R01AR048768 (NIH); NIAMS-081-1
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: Healthy adult normals
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Healthy adult participants with no history of knee injury or osteoarthritis.
  Interventions: Other: Gait analysis, knee x-ray, and knee MRI

INTERVENTIONS:
Other: Gait analysis, knee x-ray, and knee MRI — Gait analysis, knee x-rays, and knee MRIs will be done twice for each participant, 1 week apart.

SUMMARY:
The purpose of this preliminary substudy to the parent study "Aerobic Exercise Intervention for Knee Osteoarthritis" is to determine the repeatability and reproducibility of various measurement techniques.

DETAILED DESCRIPTION:
The purpose of this preliminary substudy to the parent study "Aerobic Exercise Intervention for Knee Osteoarthritis" is to determine the repeatability and reproducibility of various measurement techniques. The study will enroll healthy volunteers. All participants will receive x-rays and MRI examinations of the knees. Walking characteristics will be evaluated in a Motion Analysis Lab; this will involve taping reflective markers to participants' skin and having them walk on a level surface and up and down stairs. All participants will be evaluated two times, with a 1-week period between evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Previous knee injury, knee pain, or knee osteoarthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2002-11; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Day-to-day and inter/intra examiner repeatability of the techniques to be used in NIH grant R01 AR48768 | Measured two times, with a 1-week period between evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Kenton R. Kaufman, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Schmidt JE, Amrami KK, Manduca A, Kaufman KR. Semi-automated digital image analysis of joint space width in knee radiographs. Skeletal Radiol. 2005 Oct;34(10):639-43. doi: 10.1007/s00256-005-0908-9. Epub 2005 May 25. PMID 15915340
- [Background] Grochowski SJ, Amrami KK, Kaufman K. Semi-automated digital image analysis of patellofemoral joint space width from lateral knee radiographs. Skeletal Radiol. 2005 Oct;34(10):644-8. doi: 10.1007/s00256-005-0944-5. Epub 2005 Jul 15. PMID 16021447
- [Background] Koff MF, Amrami KK, Kaufman KR. Clinical evaluation of T2 values of patellar cartilage in patients with osteoarthritis. Osteoarthritis Cartilage. 2007 Feb;15(2):198-204. doi: 10.1016/j.joca.2006.07.007. Epub 2006 Sep 1. PMID 16949313
- [Background] Agnesi F, Amrami KK, Frigo CA, Kaufman KR. Semiautomated digital analysis of knee joint space width using MR images. Skeletal Radiol. 2007 May;36(5):437-44. doi: 10.1007/s00256-006-0245-7. Epub 2007 Jan 23. PMID 17242952